CLINICAL TRIAL: NCT02453555
Title: A Phase III, Randomised, Double-blind, Parallel Group, 52 Week Study to Evaluate Efficacy and Safety of Once Daily Empagliflozin and Linagliptin Fixed Dose Combination Compared With Linagliptin Plus Placebo in Japanese Type 2 Diabetes Mellitus Patients With Insufficient Glycaemic Control After 16 Weeks Treatment With Once Daily Linagliptin 5 mg.
Brief Title: Empagliflozin Add on to Linagliptin Study in Japanese Patient With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1275.19
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin; Tablets; empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Linagliptin (Active Comparator): patient to receive 5 mg linagliptin once daily
  Interventions: Drug: Linagliptin; Drug: Empagliflozin placebo + linagliptin placebo low dose; Drug: Empa + lina highdose placebo
- Empagliflozin + linagliptin low dose (Experimental): patient to receive one tablet once daily
  Interventions: Drug: Empagliflozin + linagliptin low dose; Drug: Linagliptin placebo
- Empagliflozin + linagliptin high dose (Experimental): patient to receive one tablet once daily
  Interventions: Drug: Linagliptin placebo; Drug: Empagliflozin + linagliptin high dose
- Linagliptin placebo (Placebo Comparator)
  Interventions: Drug: Empagliflozin + linagliptin low dose; Drug: Linagliptin placebo; Drug: Empagliflozin + linagliptin high dose
- Empagliflozin + linagliptin high dose placebo (Placebo Comparator)
  Interventions: Drug: Linagliptin; Drug: Empa + lina highdose placebo
- Empagliflozin + linagliptin low dose placebo (Placebo Comparator)
  Interventions: Drug: Linagliptin; Drug: Empagliflozin placebo + linagliptin placebo low dose

INTERVENTIONS:
Drug: Linagliptin
  Other Names: tablet
  Arms: Empagliflozin + linagliptin high dose placebo; Empagliflozin + linagliptin low dose placebo; Linagliptin
Drug: Empagliflozin placebo + linagliptin placebo low dose — Matching placebo empagliflozin + linagliptin
  Arms: Empagliflozin + linagliptin low dose placebo; Linagliptin
Drug: Empagliflozin + linagliptin low dose — tablet
  Arms: Empagliflozin + linagliptin low dose; Linagliptin placebo
Drug: Linagliptin placebo — Matching placebo linagliptin
  Arms: Empagliflozin + linagliptin high dose; Empagliflozin + linagliptin low dose; Linagliptin placebo
Drug: Empagliflozin + linagliptin high dose — tablet
  Arms: Empagliflozin + linagliptin high dose; Linagliptin placebo
Drug: Empa + lina highdose placebo
  Arms: Empagliflozin + linagliptin high dose placebo; Linagliptin

SUMMARY:
This trial will compare the use of fixed dose combination of empagliflozin and linagliptin to linagliptin alone in patient with type 2 diabetes mellitus

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of Type-2 Diabetes Mellitus (T2DM) prior to informed consent
2. Male and female patients on diet and exercise regimen for at least 12 weeks prior to informed consent who are:

   * 1 drug-naïve, defined as no antidiabetic drugs for at least 12 weeks prior to informed consent, or
   * 2 pre-treated with one oral antidiabetic drug (for sulfonylurea, with up to half of the maximum approved dose) on stable dosage for at least 12 weeks prior to informed consent (for thiazolidinedione, therapy has to be unchanged for at least 18 weeks prior to the informed consent, for linagliptin 5 mg at least 16 weeks prior to Visit 1). Individual antidiabetic drug (except linagliptin) will have to be discontinued at Visit 1.
3. HbA1c at Visit 1

   * 1 HbA1c =8.0% and =10.5% for patients who are drug-naïve, or
   * 2 HbA1c =7.5% and =10.5% for patients with one oral antidiabetic drug (except linagliptin), or
   * 3 HbA1c =7.5% and =10.0% for patients with linagliptin 5 mg
4. HbA1c =7.5% and =10.0% at Visit 4 for randomisation into the double-blind treatment period. Patient who are pre-treated with linagliptin 5 mg for 16 weeks or more prior to Visit 1 and meet the criteria of HbA1c can directly move on to the run-in (Visit 4).
5. Age =20 years at informed consent
6. BMI =40.0 kg/m2 at Visit 1 (screening)
7. Signed and dated written informed consent by date of Visit 1 in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion criteria:

1. Uncontrolled hyperglycemia with a glucose level >270 mg/dL (>15.0 mmol/L) after an overnight fast during the open-label stabilisation period (from Visit 2 to Visit 4) and run-in period (from Visit 4 to Visit 5) , confirmed by a second measurement (not on the same day and done either at the central or at local laboratory).
2. Acute coronary syndrome (ST-elevation myocardial infarction [STEMI], non-STEMI, and unstable angina pectoris), stroke or transient ischemic attack within 12 weeks prior to informed consent
3. Indication of liver disease, defined by serum levels of either alanine aminotransferase (ALT Serum glutamic pyruvate transaminase [SGPT]), aspartate aminotransferase (AST, Serum glutamic oxaloacetic transaminase [SGOT]), or alkaline phosphatase (ALP) above 3 x upper limit of normal (ULN) as determined during screening, open-label stabilisation period and/or run-in period
4. Impaired renal function, defined as estimated glomerular filtration rate (eGFR) <45 mL/min/1.73 m2 (MDRD formula) as determined during screening, open-label stabilisation period and/or run-in period
5. Known hereditary galactose intolerance
6. Known contraindications to linagliptin and empagliflozin according to the Japanese label
7. Any previous (within 2 years prior to informed consent) or planned bariatric surgery (or any other weight loss surgery) or other gastrointestinal surgery that induce chronic malabsorption
8. Medical history of cancer (except for resected non-invasive basal cell or squamous carcinoma) and/or treatment for cancer within the last 5 years
9. Known blood dyscrasias or any disorders causing haemolysis or unstable red blood cell (RBC) count (e.g. malaria, babesiosis, haemolytic anaemia).
10. Treatment with insulin, Glucagon-like peptide-1 agonists, within 12 weeks prior to informed consent
11. Treatment with anti-obesity drugs within 12 weeks prior to informed consent or any other treatment at the time of screening (i.e., surgery, aggressive diet regimen, etc.) leading to unstable body weight
12. Current treatment with systemic steroids (other than inhaled or topical steroids) at informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent or any other uncontrolled endocrine disorder except T2DM
13. Pre-menopausal women (last menstruation =1 year prior to informed consent) who:

    * 1 are nursing or pregnant or
    * 2 are of child-bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the trial and do not agree to submit to periodic pregnancy testing during participation in the trial. Acceptable methods of birth control include tubal ligation, intra uterine devices/systems, oral contraceptives, complete sexual abstinence, double barrier method and vasectomised partner
14. Known or suspected allergy or hypersensitivity to trial products or related products (e.g., Dipeptidyl-peptidase-4 inhibitors or Sodium-glucose co-transporter-2 inhibitors)
15. Alcohol or drug abuse within the 12 weeks prior to informed consent that would interfere with trial participation or any ongoing condition leading to a decreased compliance to trial procedures or trial drug intake, by the judgment of the investigator
16. Intake of an investigational drug in another trial within 30 days prior to Visit 1 or participation in the follow-up period of another trial (participation in observational studies is permitted)
17. Any other clinical condition that, in the opinion of the investigator, would jeopardize patient's safety while participating in this clinical trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2015-05-14 (Actual); Primary Completion 2016-08-26 (Actual); Study Completion 2017-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (40):
- Japan (40):
  - Nagoya Kyoritsu Hospital, Aichi, Nagoya
  - Kashiwa City Hospital, Chiba, Kashiwa
  - Otabe internal medicine clinic, Fukuoka, Fukuoka
  - Nakamura Cardiovascular Clinic, Fukuoka, Itoshima
  - Tanaka I.M. Clinic, Fukuoka, I.M., Fukuoka, Kurume
  - Seino I.M. Clinic, Fukushima, I.M., Fukushima, Koriyama
  - Hiraoka Naika Clinic, Hiroshima, I.M., Hiroshima, Hiroshima
  - Matsuda Cardiovascular Clinic, Hokkaido, Sapporo
  - Teine Keijinkai Clinic, Hokkaido, Sapporo
  - Mita Internal Medicine Cardiology Clinic, Hokkaido, Sapporo
  - Miyanosawa Clinic of Internal Medicine and Cardiology, Hokkaido, Sapporo
  - Itabashi Diabetic medicine and Dermatology Clinic, Ibaraki, Koga
  - Nakakinen Clinic, Ibaraki, Naka
  - Kubota Clinic, Kanagawa, Kawasaki
  - Kitasato University Hospital, Kanagawa, Sagamihara
  - H.E.C Science Clinic, Kanagawa, Yokohama
  - Yoshimasa Diabetes & Endocrine Clinic, Kyoto, Kyoto
  - Rakuwakai Otowa Hospital, Kyoto, Kyoto
  - Medical Corporation Hayashi Katagihara Clinic, Kyoto, Kyoto
  - Miyamoto Naika Clinic, Nagano, I.M., Nagano, Matsumoto
  - Gibo Hepatology Clinic, Nagano, Digestive Tract I.M., Nagano, Matsumoto
  - Takekawa Clinic, Osaka, I.M., Osaka, Higashi-Osaka
  - Medical Corporation Koseikai Fukuda Naika Clinic, Osaka, Osaka
  - Kinugawa Cardiovascular Internal Medicine clinic, Osaka, Osaka
  - Sato Hospital, Osaka, Osaka
  - Nakaoka Clinic, Osaka, Osaka
  - OCROM Clinic, Osaka, Suita
  - Miyauchi Medical Center, Osaka, Takatsuki
  - Medical Corporation Shinseikai Mashiba Clinic, Saitama, Hanno
  - Asano Clinic, Saitama, Kawagoe
  - Medical Corporation Fusa Shimizu Clinic Fusa, Saitama, Saitama
  - Ogino Clinic, Saitama, Tokorozawa
  - Kanda Clinic, Tokyo, Chiyoda-ku
  - Fukuwa Clinic, Tokyo, Chuo-ku
  - Tokyo-Eki Center-building Clinic, Tokyo, Chuo-ku
  - Myojin Tou Clinic, Tokyo, Hachioji
  - Sawai Medical Clinic, Tokyo, Koto-ku
  - Mishuku Hospital, Tokyo, Meguro-ku
  - Toshiba General Hospital, Tokyo, Shinagawa-ku
  - ToCROM Clinic, Tokyo, Shinjuku-ku

REFERENCES:
- [Derived] Kawamori R, Haneda M, Suzaki K, Cheng G, Shiki K, Miyamoto Y, Solimando F, Lee C, Lee J, George J. Empagliflozin as add-on to linagliptin in a fixed-dose combination in Japanese patients with type 2 diabetes: Glycaemic efficacy and safety profile in a 52-week, randomized, placebo-controlled trial. Diabetes Obes Metab. 2018 Sep;20(9):2200-2209. doi: 10.1111/dom.13352. Epub 2018 Jun 1. PMID 29766636

RESULTS

PARTICIPANT FLOW:
Groups:
- Empagliflozin 10 Milligram (mg)/Linagliptin 5 Milligram (mg): Patients were administered a fixed dose combination (FDC) of 10 mg Empagliflozin and 5 mg Linagliptin tablet along with matching placebo of Linagliptin 5 mg orally once daily for 24 weeks of double-blind treatment period.
- Linagliptin 5 mg + Placebo 10 mg: Patients were administered a matching placebo of FDC of 10 mg Empagliflozin and 5 mg Linagliptin tablet along with Linagliptin 5 mg orally once daily for 24 weeks of double-blind treatment period.
- Empagliflozin 25 mg/Linagliptin 5 mg (Extension Period): Patients with insufficient response based on Glycosylated haemoglobin A1c (HbA1c) after 24-week of double-blind treatment period were up-titrated to a FDC of 25 mg Empagliflozin and 5 mg Linagliptin tablet along with matching placebo of Linagliptin 5 mg orally once daily for 24 weeks of up-titration period (from Week 28 to Week 52).
- Empagliflozin 10 mg/Linagliptin 5 mg (Extension Period): Patients with sufficient response based on HbA1c after 24-week of double-blind treatment period were continued on a FDC of 10 mg Empagliflozin and 5 mg Linagliptin tablet along with matching placebo of Linagliptin 5 mg orally once daily for subsequent 28 weeks of extension period.
- Linagliptin 5 mg + Placebo 25 mg (Extension Period): Patients with insufficient response based on HbA1c after 24-week of double-blind treatment period were up-titrated to receive a matching placebo of FDC of 25 mg Empagliflozin and 5 mg Linagliptin tablet along with Linagliptin 5 mg orally once daily for 24 weeks of up-titration period (from Week 28 to Week 52).
- Linagliptin 5 mg + Placebo 10 mg (Extension Period): Patients with sufficient response based on HbA1c after 24-week of double-blind treatment period were continued on a matching placebo of FDC of 10 mg Empagliflozin and 5 mg Linagliptin tablet along with Linagliptin 5 mg orally once daily for subsequent 28 weeks of extension period.
Period: 24-week Double-blind Treatment Period
Arm/Group | Empagliflozin 10 Milligram (mg)/Linagliptin 5 Milligram (mg) | Linagliptin 5 mg + Placebo 10 mg | Empagliflozin 25 mg/Linagliptin 5 mg (Extension Period) | Empagliflozin 10 mg/Linagliptin 5 mg (Extension Period) | Linagliptin 5 mg + Placebo 25 mg (Extension Period) | Linagliptin 5 mg + Placebo 10 mg (Extension Period)
Started | 182 (Started are treated subjects.) | 93 (Started are treated subjects.) | 0 (This reporting group is not applicable in this period.) | 0 (This reporting group is not applicable in this period.) | 0 (This reporting group is not applicable in this period.) | 0 (This reporting group is not applicable in this period.)
Completed | 177 | 86 | 0 | 0 | 0 | 0
Not Completed | 5 | 7 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 0 | 0 | 0 | 0
Not completed — Other than specified above | 0 | 3 | 0 | 0 | 0 | 0
Period: Extension Period
Arm/Group | Empagliflozin 10 Milligram (mg)/Linagliptin 5 Milligram (mg) | Linagliptin 5 mg + Placebo 10 mg | Empagliflozin 25 mg/Linagliptin 5 mg (Extension Period) | Empagliflozin 10 mg/Linagliptin 5 mg (Extension Period) | Linagliptin 5 mg + Placebo 25 mg (Extension Period) | Linagliptin 5 mg + Placebo 10 mg (Extension Period)
Started | 0 (This reporting group is not applicable in this period.) | 0 (This reporting group is not applicable in this period.) | 126 | 51 | 80 | 6
Completed | 0 | 0 | 123 | 49 | 79 | 5
Not Completed | 0 | 0 | 3 | 2 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 2 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) consisted of all patients who were randomised and treated with at least 1 dose of trial drug and had a baseline HbA1c assessment and at least 1 on-treatment HbA1c assessment during the 24 week double-blind part of the trial.
Groups:
- Empagliflozin 10 mg/Linagliptin 5 mg: Patients were administered a fixed dose combination (FDC) of 10 mg Empagliflozin and 5 mg Linagliptin tablet along with matching placebo of Linagliptin 5 mg orally once daily for 24 weeks of double-blind treatment period.
- Total: Total of all reporting groups
Arm/Group | Empagliflozin 10 mg/Linagliptin 5 mg | Linagliptin 5 mg + Placebo 10 mg | Total
Number analyzed (Participants) | 182 | 93 | 275
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.0 (9.9) | 59.8 (10.8) | 59.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 21 | 61
  Male | 142 | 72 | 214

OUTCOME MEASURES:

1. Primary Outcome: Change of Glycosylated Haemoglobin A1c (Glycosylated Haemoglobin A1c After 24 Weeks of Double-blind Treatment From Baseline)
Description: Change from baseline in Glycosylated haemoglobin A1c (HbA1c) at Week 24 was calculated as: HbA1c at Week 24 - HbA1c at baseline. Baseline is referred to the last observed measurement prior to the administration of randomized trial medication. Adjusted mean (Least square mean) and its standard error (SE) is presented.
Time Frame: Baseline and 24 week
Population: The primary analysis was performed on the FAS (observed case [OC]) with treatment assignment as randomised.
Measure: Least Squares Mean (Standard Error); unit: Percentage (%)
Arm/Group | Empagliflozin 10 mg/Linagliptin 5 mg | Linagliptin 5 mg + Placebo 10 mg
Number analyzed (Participants) | 182 | 93
Percentage (%) | -0.93 (0.06) | 0.21 (0.09)
Statistical Analysis 1: Comparison: Empagliflozin 10 mg/Linagliptin 5 mg vs Linagliptin 5 mg + Placebo 10 mg; A restricted maximum likelihood (REML)-based mixed model repeated measures (MMRM) approach was used with baseline HbA1c as linear covariate and baseline estimated glomerular filtration rate (eGFR) (Modification of Diet in Renal Disease [MDRD] formula), prior use of antidiabetic drug, treatment, visit, visit by Treatment interaction as fixed effect(s). The covariance used to fit the model was unstructured; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted Mean Difference (Net) = -1.14, 95% CI 2-sided [-1.36 to -0.91], Standard Error of Mean 0.11 — Adjusted Mean Difference was calculated as: (adjusted mean change from baseline in HbA1c at Week 24 in Empagliflozin 10 mg/linagliptin 5 mg group) - (adjusted mean change from baseline in HbA1c at Week 24 in Linagliptin 5 mg + Placebo 10 mg group)

2. Secondary Outcome: Change in HbA1c From Week 28 at Week 52 (Empagliflozin 25 mg/Linagliptin 5 mg Only)
Description: Change from Week 28 in HbA1c at Week 52 was calculated as: HbA1c at Week 52 - HbA1c at Week 28. Week 28 (pre up-titration) is referred to the last observed measurement prior to the first administration of any double-blind randomized trial medication in the up-titration period. Adjusted mean (Least square mean) and its standard error (SE) is presented.
  This endpoint was based on 1 group of the Full analysis set with up-titration (FASUT-II) whose dose was up-titrated to Empagliflozin 25 mg/Linagliptin 5 mg fixed dose combination thus there is no comparison group. Hence, no comparison is made. A restricted maximum likelihood (REML)-based mixed model repeated measures (MMRM) approach was used with baseline HbA1c as linear covariate and baseline eGFR, prior use of antidiabetic drug, visit as fixed effect(s). The covariance used to fit the model was unstructured.
Time Frame: 28 Week (pre up-titration) and 52 Week
Population: The full analysis set with up-titration-I (FASUT-I) consisted of all patients who were up-titrated and were treated with at least 1 dose of Empagliflozin 25 mg/linagliptin 5 mg or Linagliptin 5 mg + Placebo 25 mg after dose up-titration and who had a baseline HbA1c assessment and at least 1 on-treatment HbA1c assessment after dose up-titration.
Measure: Least Squares Mean (Standard Error); unit: Percentage (%)
Groups:
- Empagliflozin 25 mg/Linagliptin 5 mg: Patients with insufficient response based on HbA1c after 24-week of double-blind treatment period were up-titrated to a FDC of 25 mg Empagliflozin and 5 mg Linagliptin tablet along with matching placebo of Linagliptin 5 mg orally once daily for 24 weeks of up-titration period (from Week 28 to Week 52).
Arm/Group | Empagliflozin 25 mg/Linagliptin 5 mg
Number analyzed (Participants) | 124
Percentage (%) | -0.21 (0.03)

3. Secondary Outcome: Change in HbA1c From Baseline at Week 52 (All Empagliflozin Versus All Placebo)
Description: Change from baseline in HbA1c at Week 52 was calculated as: HbA1c at Week 52 - HbA1c at baseline. Baseline is referred to the last observed measurement prior to the administration of randomized trial medication. Adjusted mean (Least square mean) and its standard error (SE) is presented.
Time Frame: Baseline and 52 week
Population: The analysis was performed on the FAS (observed case [OC]) with treatment assignment as randomised.
Measure: Least Squares Mean (Standard Error); unit: Percentage (%)
Groups:
- All Empagliflozin: Patients were administered a FDC of 10 mg Empagliflozin and 5 mg Linagliptin tablet along with matching placebo of Linagliptin 5 mg orally once daily for 24 weeks of double-blind treatment period. In the up-titration period (from Week 28 to Week 52), patients with insufficient response measured after 24 weeks of double-blind treatment got up-titrated to FDC of 25 mg Empagliflozin and 5 mg Linagliptin while the other patients kept the same dose.
- All Placebo: Patients were administered a matching placebo of FDC of 10 mg Empagliflozin and 5 mg Linagliptin tablet along with Linagliptin 5 mg orally once daily for 24 weeks of double-blind treatment period. In the up-titration period (from Week 28 to Week 52), patients with insufficient response measured after 24 weeks of double-blind treatment got up-titrated to matching placebo of FDC of 25 mg Empagliflozin and 5 mg Linagliptin while the other patients kept the same dose.
Arm/Group | All Empagliflozin | All Placebo
Number analyzed (Participants) | 182 | 93
Percentage (%) | -1.16 (0.06) | 0.06 (0.10)
Statistical Analysis 1: Comparison: All Empagliflozin vs All Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted Mean Difference (Net) = -1.22, 95% CI 2-sided [-1.45 to -0.99], Standard Error of Mean 0.12 — Adjusted Mean Difference was calculated as: (adjusted mean change from baseline in HbA1c at Week 52 in All Empagliflozin group) - (adjusted mean change from baseline in HbA1c at Week 52 in All Placebo group)

4. Secondary Outcome: Change in HbA1c From Baseline at Week 52 (Empagliflozin 25 mg/Linagliptin 5 mg Versus Linagliptin 5 mg + Placebo 25 mg)
Description: as for outcome 3
Time Frame: Baseline and 52 week
Population: FASUT-I
Measure: Least Squares Mean (Standard Error); unit: Percentage (%)
Groups:
- Linagliptin 5 mg + Placebo 25 mg: Patients with insufficient response based on HbA1c after 24-week of double-blind treatment period were up-titrated to receive a matching placebo of FDC of 25 mg Empagliflozin and 5 mg Linagliptin tablet along with Linagliptin 5 mg orally once daily for 24 weeks of up-titration period (from Week 28 to Week 52).
Arm/Group | Empagliflozin 25 mg/Linagliptin 5 mg | Linagliptin 5 mg + Placebo 25 mg
Number analyzed (Participants) | 126 | 80
Percentage (%) | -1.10 (0.07) | 0.11 (0.10)
Statistical Analysis 1: Comparison: Empagliflozin 25 mg/Linagliptin 5 mg vs Linagliptin 5 mg + Placebo 25 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted Mean Difference (Net) = -1.21, 95% CI 2-sided [-1.45 to -0.96], Standard Error of Mean 0.12 — Adjusted Mean Difference was calculated as: (adjusted mean change from baseline in HbA1c at Week 52 in Empagliflozin 25 mg/linagliptin 5 mg group) - (adjusted mean change from baseline in HbA1c at Week 52 in Linagliptin 5 mg + Placebo 25 mg group)

5. Secondary Outcome: Change in HbA1c From Baseline at Week 52 (Empagliflozin 25 mg/Linagliptin 5 mg Versus All Placebo)
Description: as for outcome 3
Time Frame: Baseline and 52 week
Population: Full analysis set with up-titration-II consisted patients who were up-titrated to Empagliflozin 25/linagliptin 5 and were treated with at least 1 dose after dose up-titration and who were randomized to receive Linagliptin 5 + Placebo 10 or Linagliptin 5 + Placebo 25 and who had HbA1c assessment at baseline and at least once after dose up-titration.
Measure: Least Squares Mean (Standard Error); unit: Percentage (%)
Arm/Group | Empagliflozin 25 mg/Linagliptin 5 mg | All Placebo
Number analyzed (Participants) | 126 | 86
Percentage (%) | -1.10 (0.07) | -0.01 (0.10)
Statistical Analysis 1: Comparison: Empagliflozin 25 mg/Linagliptin 5 mg vs All Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted Mean Difference (Net) = -1.09, 95% CI 2-sided [-1.34 to -0.84], Standard Error of Mean 0.13 — Adjusted Mean Difference was calculated as: (adjusted mean change from baseline in HbA1c at Week 52 in Empagliflozin 25 mg/linagliptin 5 mg group) - (adjusted mean change from baseline in HbA1c at Week 52 in All Placebo group)

ADVERSE EVENTS:
Time Frame: From first drug administration till 52 weeks, up to 7 days after last drug administration.
Description: TreatedSet(TS) included of patients who were randomised and treated with at least 1Dose of trial drug. Patients were randomized into 2Groups and remained in these groups after 28Weeks treatment. Patients got dose up-titrated after treatment,but had the same medication as it was before up-titrated.Data was reported for 2Arms based on randomization.
Arm/Group | All Empagliflozin | All Placebo
Serious Adverse Events (participants affected / at risk) | 8/182 | 1/93
Other Adverse Events (participants affected / at risk) | 62/182 | 46/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Empagliflozin (N=182) | All Placebo (N=93)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Prinzmetal angina (Cardiac disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Empagliflozin (N=182) | All Placebo (N=93)
Nasopharyngitis (Infections and infestations) | 35 | 34
Asymptomatic bacteriuria (Infections and infestations) | 13 | 6
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 14 | 10
Blood ketone body increased (Investigations) | 12 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.